CLINICAL TRIAL: NCT00388115
Title: A Pilot Study of Radiofrequency Ablation of Early Invasive and In Situ Breast Cancer
Brief Title: Radiofrequency Ablation in Treating Patients With Early Invasive Breast Cancer or Ductal Carcinoma in Situ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Vijay Khatri, MD, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000505536; P30CA093373 (NIH); UCD-123 (Other: University of California, Davis - Cancer Center); UCD-200210277-6 (Other: University of California, Davis - IRB)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-03

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ; stage I breast cancer; stage II breast cancer; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Neoadjuvant Therapy; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RFA prior to surgery (Experimental)
  Interventions: Procedure: conventional surgery; Procedure: neoadjuvant therapy; Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: conventional surgery — Standard of care lumpectomy or mastectomy following RFA
Procedure: neoadjuvant therapy — Standard of care lumpectomy or mastectomy following RFA
Procedure: radiofrequency ablation — A small diameter needle is inserted through the skin and directly into the tumor for the purpose of supplying RF current. Initial power of the RF generator will start at 5-10 watts. The power will increase by 5-10 watts every minute until impedance of the system automatically stops the RF treatment.
  Other Names: RFA

SUMMARY:
RATIONALE: Radiofrequency ablation uses a high-frequency, electric current to kill tumor cells. Giving radiofrequency ablation before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This clinical trial is studying how well radiofrequency ablation followed by surgery works in treating patients with early invasive breast cancer or ductal carcinoma in situ.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effectiveness of radiofrequency ablation (RFA), in terms of amount of tumor coagulated and viable cell count, in patients with early invasive breast cancer or low- or intermediate-grade ductal carcinoma in situ.

Secondary

* Determine the size, configuration, and pathological features of human breast tumors after treatment with RFA.
* Determine whether RFA energy applied to breast cancer will result in cancer cell death.
* Determine whether tumor-free margins are achieved by RFA in these patients.
* Determine the rate of acute toxicities to skin after surgery in patients treated with this regimen.

OUTLINE: This is a pilot study.

* Pre-radiofrequency ablation (RFA) procedures: Patients undergo staging by MRI assessment to determine the size of their tumor. Patients with nonpalpable lesions must undergo placement of a metallic clip in the center of their tumor and a hook wire to guide surgical excision by intraoperative ultrasound imaging. Patients with invasive breast cancer undergo axillary lymph node dissection or sentinel lymph node biopsy (SLNB) for axillary lymph node staging. Patients with ductal carcinoma in situ proceed directly to RFA/resection since they do not require axillary staging.
* RFA: Patients undergo RFA comprising insertion of a multiple-needle electrode into the breast tumor under direct guidance of ultrasonography and the metallic clip placed preoperatively in the lesion.
* Surgical resection of RFA area: After RFA is completed, the electrode is removed and patients undergo wide local excision of the residual tumor or mastectomy.

After completion of study therapy, patients are followed periodically for up to 4 months.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Females of ages ≥18 years.
* Core biopsy proven invasive breast cancer OR
* Core biopsy proven low or intermediate grade DCIS.
* Tumor less than or equal to 2.0 cm in diameter.
* No prior surgical treatment for breast cancer within 30 days.
* Life expectancy of > 10 years, not including the diagnosis of cancer.
* ECOG performance status of 0-2.
* Informed consent given.
* Multifocal invasive breast cancer patients are eligible. All tumors that are palpable or visualized by USS can be treated.

Exclusion Criteria:

* Male subjects.
* Ages < 18 years.
* Breast tumor > 2.0 cm in diameter.
* Evidence of distant metastatic disease.
* Evidence of diffuse calcification suggestive of extensive or multifocal DCIS.
* High grade DCIS or presence of comedo-necrosis because these lesions can be associated with invasive breast cancer, which would go undetected if the lesion is entirely destroyed by the RF ablation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2001-10; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Number and proportion of patients with viable cancer cells remaining in the resected specimen as measured by enzyme cell viability analysis and amount of tumor coagulated at post-treatment biopsy | At completion of study

SECONDARY OUTCOMES:
Number and proportion of patients with uncoagulated tumor remnant at post-treatment biopsy | At completion of study
Number and proportion of patients with and without tumor in the margin | At completion of study
Rate of acute skin toxicity | At completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Khatri, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States